CLINICAL TRIAL: NCT02797990
Title: Mother vs. Child? Healthcare Worker Perceptions of Conflict Between Maternal Autonomy and Child Health When Providing Care for Pregnant Women Engaging in Problematic Substance Use
Brief Title: Conflict Between Maternal Autonomy and Child Health in Substance-use
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 10890; 201264 (Other: IRAS Number); FI0816115 (Other: LSHTM Sponsorship Certification Number)
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-05

CONDITIONS: Substance-Related Disorders; Alcohol-Related Disorders; Amphetamine-Related Disorders; Inhalant Abuse; Cocaine-Related Disorders; Opioid-Related Disorders; Marijuana Abuse; Substance Abuse, Intravenous; Neonatal Abstinence Syndrome; Pregnancy; Pregnancy, High-Risk
Keywords: [G08.686.785.760.769.500]; [G08.686.785.760.769]; [N02.360]; [C25.775.650]; [C25.775.793]; [C25.775.635]; [C25.775.675]; [C25.775.300]; [C25.775.467]; [C25.775.225]; [C25.775.100]; [C25.775]
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders; Amphetamine-Related Disorders; Inhalant Abuse; Cocaine-Related Disorders; Opioid-Related Disorders; Marijuana Abuse; Substance Abuse, Intravenous; Neonatal Abstinence Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Qualitative project, comprising open-ended semi-structured interviews with healthcare workers, who provide antenatal care to substance-using women.

DETAILED DESCRIPTION:
Maternal substance use during pregnancy (including legal and illicit substances) is a fairly common global phenomenon, including in the UK. This can have significant effects on pregnancy, infant outcome and enduring consequences into adolescence. Babies born with neonatal abstinence syndrome may spend months in neonatal care units, requiring complex, 24hour care. Here, healthcare workers may experience conflict between preserving maternal autonomy, and the challenge of caring for a withdrawing newborn.

However, there is discrepancy between the objectives of policy-makers "Reducing the harm to children from parental problem drug use should become a main objective of policy and practice" and those recommended in healthcare "These women need supportive and coordinated care during pregnancy." Therefore, conflict arises between mother-centred and child-centred models of caring for pregnant women who use substances.

The objective of the proposed project is to investigate how healthcare workers providing treatment for pregnant women who use illicit substances perceive their duty of care and whether they experience tension between the conflicting objectives of mother-centred and child-centred approaches through semi-structured qualitative interviews. The investigators will explore the ways in which healthcare workers frame problematic substance misuse in pregnant women, what they perceive to be the major challenges in providing care and their views on the responsibility of a mother to have a healthy baby. The main hypothesis is that healthcare workers providing care for pregnant women engaging in problematic substance misuse experience conflict between mother-centred and child- centred approaches to care.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers will be recruited based on their employment status; they must currently provide some form of antenatal are for women who engage in problematic use of substances (limited to illicit drugs, excluding tobacco and alcohol).
* Healthcare workers will not be restricted by age, and all genders will be included. As the research is qualitative, a representative same is unnecessary.

Exclusion Criteria:

* Healthcare workers will be excluded if they do not have experience of providing ante-natal care for women who engage in problematic substance misuse (limited to illicit drugs, excluding tobacco and alcohol) during their pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare workers may include Specialist Midwives, Obstetricians, Substance Misuse Charge Nurses, Neonatologists and Health Visitors. Women using substances are defined as those who are being seen at the clinic (either due to self-referral, or due to referral by a healthcare worker), at any time during their pregnancy. I have personal experience of working in this clinic, which is run in an NHS hospital on the South Coast of the UK.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Perceptions of conflict between maternal and child-centred approaches | 4 months
  Qualitative data of perceptions of conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Knox, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Trevor Mann Baby Unit, Royal Sussex County Hospital, Brighton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanaullah F, Gillian M, Lavin T. Screening of substance misuse during early pregnancy in Blyth: an anonymous unlinked study. J Obstet Gynaecol. 2006 Apr;26(3):187-90. doi: 10.1080/01443610500508121. PMID 16698620